CLINICAL TRIAL: NCT02837757
Title: Everolimus Modulation of Anti-tumor T CD4 Immune Responses
Acronym: EMIR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty of patient recruitment
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: API/2014/48
Record Dates: First submitted 2016-07-13; First posted 2016-07-20 (Estimated); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Metastatic Renal Cancer
MeSH Terms: conditions — Kidney Neoplasms

ARMS (1):
- Biological samples (Experimental): Blood samples will be realized specifically to the study at inclusion (baseline before starting everolimus treatment), and then 3 months and 9 months (or at disease progression if occurs first) after initiation of everolimus treatment Peripheral blood mononuclear cell (PBMC) and serum will be collected.
  Available tumor tissues samples will be collected.
  Interventions: Other: Biological samples

INTERVENTIONS:
Other: Biological samples — blood and tumor tissue samples

SUMMARY:
Everolimus is an inhibitor of mammalian target of rapamycin, approved in patients with metastatic renal cell carcinoma.

The objective of this study is to investigated the influence of everolimus immune modulation on antitumor efficacy .

ELIGIBILITY:
Inclusion Criteria:

* Performance status ECOG-WHO 0, 1 or 2
* Metastatic renal cancer
* Patient candidate to everolimus treatment
* signed written informed consent
* fertile women with adequate contraception during the study and until 8 weeks after stopping treatment

Exclusion Criteria:

* Patients under chronic treatment with systemic corticoids or other immunosuppressive drugs (prednisone or prednisolone ≤ 10 mg/day is allowed)
* History of immune deficiency
* Hypersensitivity against rapamycin and derived
* Prior history of other malignancy except for: basal cell carcinoma of the skin, cervical intra-epithelial neoplasia and other cancer curatively treated with no evidence of disease for at least 5 years
* Active autoimmune diseases, HIV, hepatitis C or B virus
* Patients with any medical or psychiatric condition or disease,
* Patients under guardianship, curatorship or under the protection of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-11; Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Change in regulatory T cell counts during treatment with everolimus | 9 months after everolimus initiation

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - Hôpital Nord Franche-Comté, Montbéliard
  - Hôpital Européen Georges Pompidou, Paris